CLINICAL TRIAL: NCT05502575
Title: Everyday Stress Response Targets in the Science of Behavior Change
Brief Title: Understanding Everyday Stress
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); University of California, Merced (Other); Stony Brook University (Other); Oregon State University (Other)
Responsible Party: Principal Investigator, Joshua Smyth, Distinguished Professor, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UH3AG052167 (NIH); UH3AG052167 (NIH)
Record Dates: First submitted 2019-09-02; First posted 2022-08-16 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Stress; Psychological Stress
Keywords: Stress; Stress Management; Health Behaviors; Experimental Medicine; Science of Behavior Change
MeSH Terms: conditions — Stress, Psychological; Health Behavior

STUDY DESIGN:
Intervention Model Description: A comparative trial of two stress management approaches for the improvement of stress responses, sleep, and physical activity in everyday life.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants, research staff, and outcome assessors will be blind to condition assignment and to specific details of the intervention. Investigators will be blind to condition assignment until the conclusion of data collection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-monitoring and individualized stress management (Experimental): Self-monitoring and individualized stress management materials available on a smartphone.
  Interventions: Behavioral: Self-monitoring and personalized stress management
- Self-monitoring and general stress management (Active Comparator): Self-monitoring and general stress management materials available on a smartphone.
  Interventions: Behavioral: Self-monitoring and general stress management

INTERVENTIONS:
Behavioral: Self-monitoring and personalized stress management — Self-monitoring and personalized stress management education and materials.
  Arms: Self-monitoring and individualized stress management
Behavioral: Self-monitoring and general stress management — Self-monitoring and general stress management education and materials.
  Arms: Self-monitoring and general stress management

SUMMARY:
This research study is being done to better understand how people experience stress in everyday life and how that stress may relate to sleep and physical activity. We are also testing stress management approaches that are intended to reduce stress responses in everyday life.

DETAILED DESCRIPTION:
This research study is being done to better understand how people experience stress in everyday life and how that stress may relate to sleep and physical activity. We are also testing stress management approaches that are intended to reduce stress responses in everyday life.

This study asks participants to carry and use a study-provided smartphone to answer brief surveys during daily life for several weeks. On these surveys, participants will self-report their stress, mood, thoughts, physical activity, and sleep patterns, as well as a few other questions about where they are and what they are doing at each survey. Study participants will also wear two commercial devices on their person; one that tracks physical activity and the other sleep. Information about stress management will also be provided to participants on the study smartphone. At the end of the study, participants will be asked to return the smartphone and devices and will receive compensation for their time and effort.

The overall aim of this study is to determine the effectiveness of two stress management interventions, both delivered via the study smartphone, on the outcomes of stress responses, sleep, and physical activity.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women between the ages of 35-65 years
2. Capable of reading, understanding, and speaking English and providing written informed consent
3. Free of visual and motor impairment that would interfere with the use of a smartphone
4. In good general health, ambulatory, and free of functional activity limitations
5. Stated willingness to comply with all study procedures and availability for the duration of the study

Exclusion Criteria:

1. Diagnosed mental health condition that required a medication adjustment or hospitalization within the last 3 months
2. Primary caretaker for a parent or severely disabled child/family member
3. Inability to answer Smartphone survey messages received throughout the day due to restrictions or policies in the workplace
4. Employment that requires work between the hours of 10pm and 6am or overnight 'on-call'
5. Known allergic reactions to surgical adhesive tape
6. Self-reported or medical diagnosis of sleep apnea, score above threshold on the STOP-BANG screening, or self-reported use of a C-PAP machine
7. Inability to be physically active or who have medical contradictions for physical activity
8. Self-report of physical exercise of 200 minutes or more per week at a moderate or vigorous intensity, or 10 or more hours of walking per week
9. Use of physician prescribed sleep aids/pharmaceuticals or over the counter sleep aids for 3 or more days per week
10. Living in same household as a current or former participant
11. Unwilling to travel to the study site for in-person visits
12. Travelling for an extended period of time when scheduled for study participation or unwilling to return for in-person visit subsequently

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2023-07-14 (Actual)

PRIMARY OUTCOMES:
Stress responses in everyday life | Assessed daily for 4 weeks. Changes in stress responses from prior to intervention to during the intervention period.
  Our primary outcome assessment is psychological stress responses in everyday life. To characterize subjective stress response, we utilize brief assessments of stress response indicators that encompass three aspects of the stress response in everyday life.
  First, we assess change in subjective stress indicators from non-stressed resting state to immediately after experiencing a stressor (i.e., stress reactivity).
  Second, we assess recovery in subjective stress indicators from stress following exposure as indexed by the degree to which the individual returns to their non-stressed resting state following stress reactivity.
  Third, as stress responses may occur in isolation or repeatedly, we characterize the number of stress responses over time (the sum of observed stress response cycles in a 48-hr interval).

SECONDARY OUTCOMES:
Activity behaviors - time spent sitting | Assessed daily for 4 weeks. Changes in physical activity and sedentary behaviors from prior to intervention to during the intervention period.
  Daily number of waking minutes spent sitting, summarized as the daily average for each participant derived from an activPAL 4 accelerometer worn on the midline of the thigh.
Activity behaviors - time spent standing | Assessed daily for 4 weeks. Changes in physical activity and sedentary behaviors from prior to intervention to during the intervention period.
  Daily number of waking minutes spent standing, summarized as the daily average for each participant derived from an activPAL 4 accelerometer worn on the midline of the thigh.
Activity behaviors - time spent in light physical activity | Assessed daily for 4 weeks. Changes in physical activity and sedentary behaviors from prior to intervention to during the intervention period.
  Daily number of waking minutes spent performing light physical activity, summarized as the daily average for each participant derived from an activPAL 4 accelerometer worn on the midline of the thigh.
Activity behaviors - time spent in moderate or vigorous physical activity | Assessed daily for 4 weeks. Changes in physical activity and sedentary behaviors from prior to intervention to during the intervention period.
  Daily number of waking minutes spent performing moderate of vigorous physical activity, summarized as the daily average for each participant derived from an activPAL 4 accelerometer worn on the midline of the thigh.
Activity behaviors - total step count | Assessed daily for 4 weeks. Changes in physical activity and sedentary behaviors from prior to intervention to during the intervention period.
  Total number of daily steps taken, summarized as the daily average for each participant derived from an activPAL 4 accelerometer worn on the midline of the thigh.
Activity behaviors - total sit-stand transitions | Assessed daily for 4 weeks. Changes in physical activity and sedentary behaviors from prior to intervention to during the intervention period.
  Daily number of transitions from sitting to standing, summarized as the daily average for each participant derived from an activPAL 4 accelerometer worn on the midline of the thigh.
Activity behaviors - meets recommended moderate-vigorous activity recommendation threshold | Assessed daily for 4 weeks. Changes in physical activity and sedentary behaviors from prior to intervention to during the intervention period.
  Categorical variable denotes whether a participant achieved 21.5 minutes of MVPA on a given day (derived from a recommended weekly level MVPA is 150 minutes, transformed to compute a daily threshold of recommended MVPA).
Sleep - total sleep time | Assessed daily for 4 weeks. Changes in sleep behaviors from prior to intervention to during the intervention period.
  Total number of minutes between sleep onset and final awakening; daily total sleep time (TST) scores will be summarized as the average TST (i.e., the daily average) for each participant.
Sleep - wake after sleep onset | Assessed daily for 4 weeks. Changes in sleep behaviors from prior to intervention to during the intervention period.
  Total number of minutes that a participant spent awake between sleep onset and final awakening; daily wake after sleep onset (WASO) scores will be summarized as the average WASO (i.e., the daily average) for each participant.
Sleep - sleep efficiency | Assessed daily for 4 weeks. Changes in sleep behaviors from prior to intervention to during the intervention period.
  Daily proportion of Total Sleep Time spent in bed; daily sleep efficiency (SE) scores will be summarized as the average SE (i.e., the daily average) for each participant.
Sleep - meets recommended sleep recommendation | Assessed daily for 4 weeks. Changes in sleep behaviors from prior to intervention to during the intervention period.
  Categorical variable denotes whether a participant achieved a Total Sleep Time at least seven hours of sleep on a given day.

OTHER OUTCOMES:
Mood | Changes from baseline to post-intervention (one month later)
  12-item instrument utilizing mood items derived from the Positive and Negative Affect Schedule and Circumplex Model of Affect. Items are scored from "not at all" (10) to "extremely" (50) and combined for a score for each subscale corresponding to high and low arousal positive and negative affect (range is 30-150 on each subscale).
  High activation positive subscale: Higher scores indicate greater levels of high activation positive affect (i.e., happy, enthusiastic, excited). Low activation positive subscale: Higher scores indicate greater levels of low activation positive affect (i.e., relaxed, content, calm). High activation negative subscale: Higher scores indicate greater levels of high activation negative affect (i.e., anxious, annoyed, upset). Low activation negative subscale: Higher scores indicate greater levels of low activation negative affect (i.e., bored, sad, sluggish).
Stress | Changes from baseline to post-intervention (one month later)
  Subjective report of recent stress - 6 items assessing presence of stress in past 7 days, including global rating of overall stress, frequency, duration, stressor severity, control over the stressor, predictability, current impact of stress, thoughts about the stressor, reactivity and recovery from the stressor, and ease of recovery following the stress. Higher scores indicate higher level of recent stress.
Perceived Stress | Changes from baseline to post-intervention (one month later)
  Assessed by the Perceived Stress Scale; 14 items assessing stress in past 7 days. Items scored from "never" (10) to "very often" (50). Yields total score with all items averaged together. Minimum possible score of 10 and a maximum possible score of 50. Higher scores indicate greater levels of perceived stress
Stress-related thoughts | Changes from baseline to post-intervention (one month later)
  Perseverative cognitions measured by 5 items scored from "not at all" (0) to "very much" (100). Yields a total score reflecting the average across all items, with a range of 0-100. Higher scores reflect greater degree of perseverative cognition related to stressful topics.
Stress mindset | Changes from baseline to post-intervention (one month later)
  General stress mindset as measured by the 8-item Stress Mindset Measure. Items scored in one-unit increments with values ranging from 1 ("strongly disagree") to 5 ("strongly agree"). The scale yields a total score with all items averaged together, with a range of 1 to 5. Higher scores represent the mindset that stress is enhancing.
Social support | Changes from baseline to post-intervention (one month later)
  Social support as measured by 8-items from the Social Support Questionnaire.
  This scale has 8 items that reflect two sub-scales of 4 items each. Four items enumerate the number of people that fit the question (e.g., "In the past 30 days, how many people could you really count on to help you feel more relaxed when you were under pressure or tense?") with options ranging from 0 to 10. The remaining four items assess reported satisfaction with social support and are scored from "very dissatisfied" (0) to "very satisfied" (100). Subscale scores calculated by averaging the four-item blocks separately:
  Number subscale: higher scores indicate a greater number of people available to provide social support, with a range of 0 to 10.
  Satisfaction subscale: higher scores indicate greater levels of availability and/or satisfaction with the social support received from others, with a range of 0 to 100.
Insomnia symptoms | Changes from baseline to post-intervention (one month later)
  Insomnia symptom severity as measured using the 7-item Insomnia Severity Index.
  Items assessing difficulty falling asleep, staying asleep, and problems waking too early assessed on a scale of 0 to 4 ("none", "mild", "moderate", "severe", "very severe") with higher values indicating worse insomnia symptoms.
  Additional items assess satisfaction with sleep patterns, how noticeable sleep problems are to others, amount of worry or distress about sleep problems, and interference with daily life.
Reported sleep quality | Changes from baseline to post-intervention (one month later)
  Pittsburgh Sleep Quality Index is comprised of items that assess overall sleep quality (range "very good" to "very bad"), typical bedtime, minutes to fall asleep, wake time, total sleep time (in hours), feeling rested ("always" to "never"), frequency of medication use for sleep ("not during the last month", "less than once a week", "once or twice a week", "three or more times a week"), causes of sleep problems, and bed sharing. Each item is scored 0-3 and are used to generate a total score ranging from 0 (good sleep) to 21 (impaired sleep).
Reported physical activity | Changes from baseline to post-intervention (one month later)
  Multiple aspects of reported physical activity behavior (walking, moderate activity, vigorous activity, sedentary time, and total activity) are assessed using the International Physical Activity Questionnaire - Short Form. Units of measure are median metabolic equivalent of task (MET) minutes.
  Walking (2 items; range 0 to 33264). Higher values reflect greater durations of time reported spent walking.
  Moderate intensity activity (2 items; range 0 to 40320). Higher values reflect greater moderate-intensity physical activity.
  Vigorous intensity activity (2 items; range 0 to 80640). Higher values reflect greater vigorous-intensity physical activity.
  Total activity (6 items; range 0 to 80640). Total METs = walking METs + moderate-intensity METs + vigorous-intensity METs. Higher values reflect greater intensity-based physical activity.
  Sedentary time (2 items; range 0 to 1440). Units of measure are minutes. Higher values reflect greater sedentary time.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua M Smyth, PhD, Principal Investigator — Penn State University; Jillian A Johnson, PhD, Study Director — Penn State University
Locations (1):
- Stress, Health, and Daily Experiences Laboratory, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All available, fully deidentified, IPD will be made available for research (non-commercial) purposes two years subsequent to the conclusion of the trial.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Fully deidentified data will be made available for research (non-commercial) purposes two years subsequent to the conclusion of the trial. Data will be available for a minimum of five years, although efforts will be made to keep it available as long as possible.
Access Criteria: Non-commercial research purposes only. Data must be requested and cited appropriately.

REFERENCES:
- [Derived] Johnson JA, Zawadzki MJ, Sliwinski MJ, Almeida DM, Buxton OM, Conroy DE, Marcusson-Clavertz D, Kim J, Stawski RS, Scott SB, Sciamanna CN, Green PA, Repka EM, Toledo MJL, Sturges NL, Smyth JM. Adaptive Just-in-Time Intervention to Reduce Everyday Stress Responses: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Jan 22;14:e58985. doi: 10.2196/58985. PMID 39842791